CLINICAL TRIAL: NCT03192280
Title: Skin IaM: An Exploratory Clinical Trial to Evaluate Changes in Skin Appearance, Colour, and/or Texture Following the Induction of a Local Inflammatory Skin Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LHUB-001
Record Dates: First submitted 2017-06-16; First posted 2017-06-20 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2017-07

CONDITIONS: Skin Inflammation
MeSH Terms: conditions — Dermatitis | interventions — Leukotriene B4

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- All study participants (Experimental): Each subject will receive single topical induction application of Leukotriene B4 (LTB4) on the inner arm.
  Images of the treated area will be captured using multiple medical devices.
  Interventions: Drug: Leukotriene B4; Device: FLIR One; Device: SCIO; Device: MS Band 2; Device: AGE reader; Device: HSI prototype (PARC) hyper-spectral camera; Device: iPhone 7

INTERVENTIONS:
Drug: Leukotriene B4 — Leukotriene B4 (LTB4)
Device: FLIR One — Thermal imaging attachment to iPhone
Device: SCIO — Handheld near-IR molecular spectroscopy device
Device: MS Band 2 — Wearable "watch-like" device with multiple sensors
Device: AGE reader — Portable bench top device for in-clinic near UV assessment
Device: HSI prototype (PARC) hyper-spectral camera — Portable bench top device for in-clinic multispectral imaging
Device: iPhone 7 — Smart phone

SUMMARY:
This trial will test the feasibility of various imaging devices to detect local skin inflammation prior to clinical manifestation.

ELIGIBILITY:
Inclusion Criteria:

* Male aged >25- <40 years.
* Healthy, non-smoker.
* In the opinion of the investigator, the subject will be able to comply with the requirements of the protocol, including ability to present for all required visits.
* Subject is capable of understanding and signing an informed consent form.
* White origin (limit Skin Fitzpatrick I to III).

Exclusion Criteria:

* Male aged < 25 years or >40 years.
* Female of any age.
* Tattoos on or within 5 cm of the area to be assessed.
* Scars on or with 5 cm of the area to be assessed.
* Current, active inflammatory skin disease, or past history of any inflammatory skin disease (other than acne) such as psoriasis, atopic dermatitis.
* Suffered from any significant allergies (i.e. food, environmental, contact).
* Subjects who are immunocompromised (i.e. HIV positive, Hepatitis C, transplant, etc.), based on clinical history.
* Subjects who currently have an activated immune system (e.g from current infection or recent vaccination).
* Subjects who have a history of chronic disease such as diabetes.
* Use of investigational therapy in the preceding month prior to screening visit.
* Use of G-CSF, GM-CSF, IL-2, IFNs, erythropoietin, systemic or inhaled steroids within one month of the screening visit.
* Use of oral analgesics/anti-inflammatories (e.g. paracetamol, ibuprofen, aspirin, codeine) or topical anti-inflammatories (e.g., ibuprofen) within 5 days of the screening visit.
* Concurrent disease or conditions that may present a risk to the subjects.

Ages: 25 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2017-07-06 (Actual); Study Completion 2017-07-06 (Actual)

PRIMARY OUTCOMES:
Time-point of change from baseline and comparator in electro-magnetic spectra as measured by HSI PARC | Day 1 to Day 3
  Spectra from 400 - 1000 nm in 5 nm increments

CONTACTS AND LOCATIONS:
Overall Officials: Paul Griffin, MD, Principal Investigator — Q-Pharm Pty Limited
Locations (1):
- Investigational Site, Herston, Australia

IPD SHARING:
Plan to Share IPD: No